CLINICAL TRIAL: NCT00764816
Title: Effect of Dietary Protein Source on Phosphaturia, PTH and FGF23 in Patients With CKD 3 and 4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sharon M. Moe, MD, Indiana University Department of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0807-03
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease, stages 3 and 4; phosphaturia; phosphorus; PTH; FGF23; Dietary protein source
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypophosphatemia, Familial | interventions — Edible Grain; Caseins; Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 grain (soy) protein diet: (Active Comparator): The patient is to eat a grain (soy) protein diet for 7 days. The food is prepared by a registered dietitian.
  Interventions: Other: grain (soy) protein diet
- 2 casein (meat) protein diet (Active Comparator): The patient is to eat a casein (meat) protein diet for 7 days. The food is prepared by a registered dietitian.
  Interventions: Other: casein (meat) protein diet

INTERVENTIONS:
Other: grain (soy) protein diet — The patient is to eat a grain (soy) protein diet for 7 days. The food is prepared by a registered dietitian.
  Arms: 1 grain (soy) protein diet:
Other: casein (meat) protein diet — The patient is to eat a casein (meat) protein diet for 7 days. The food is prepared by a registered dietitian.
  Arms: 2 casein (meat) protein diet

SUMMARY:
Phosphorus is a substance in the blood that comes from food and is normally cleared from the body by the kidneys. In patients with kidney disease, excess phosphorus may build up in the body as you eat. This leads to problems with bones and blood vessels over time. In this study, we will compare the blood and urine before and after eating one week of a diet with a protein from plants (soy and grains) and before and after another one week of diet with protein from animals (meat and dairy products). The amount of phosphorus that the kidney puts out in the urine, and the changes in blood hormones in response to the diet will be measured at the beginning and end of each week on the two diets.

DETAILED DESCRIPTION:
Chronic Kidney Disease-Mineral Bone disorder (CKD-MBD) is a constellation of problems related to alterations in mineral and bone homeostasis that occur in CKD stage 3-5D (estimated GFR 60-15 ml/min). The damaged kidney is unable to fully excrete a phosphorus load, leading to a compensatory secondary hyperparathyroidism to attempt to increase urinary phosphorus excretion in order to maintain serum phosphorus in the normal range. Eventually this compensation of elevated PTH becomes pathologic and leads to abnormalities in biochemistries, bone and vascular disease, all of which are associated with morbidity and mortality in patients with CKD. Prevention of these complications is key to improved patient outcomes. Unfortunately, this normal or high normal phosphorus does not reflect the "behind the scenes" appropriate and inappropriate compensation. The use of medication to bind phosphorus from food (phosphate binders) may prevent absorption of phosphorus across the intestine and prevent or change the elevations in PTH and other hormones like FGF23. Thus, either urinary excretion of phosphorus, or changes in hormone may be more appropriate end points to evaluate efficacy of phosphate binders than is serum phosphorus.

In healthy individuals, there is variation throughout the day (diurnal) in serum phosphorus and urine phosphorus excretion, but in dialysis patients, this variability appears to be lost. No data exists for patients with stage 3 and 4 (pre-dialysis) CKD. Intestinal phosphorus absorption is also dependent on bioavailability (amount of free phosphorus available to be absorbed), which differs depending on the protein source, as the phosphorus in grain/soy diets is less bioavailable than that from protein from animal/casein protein source. In our animal model of CKD, these differences in bioavailability impact urinary phosphorus excretion and serum levels of FGF-23, but not PTH. As phosphaturia, PTH, and FGF23 may become important end points for future clinical trials, understanding diurnal variability and the relationship to diet in patients with CKD 3 and 4 with normal serum phosphorus levels is critical. We hypothesize that dietary protein source will affect the hormonal response and diurnal phosphorus homeostasis in advanced CKD. To test this hypothesis, we will examine the following specific aims in a population of CKD stage 3 and 4 subjects from the Indiana University Affiliated Nephrology Clinics and determine

1. if the dietary protein source affects fasting serum and urinary phosphorus excretion
2. if the protein source affects post prandial changes in serum and urinary phosphorus in patients
3. if changes in plasma FGF23 and PTH correlate with urinary phosphorus excretion in response to different protein sources.

We will conduct a cross over study to assess blood and urine after one week of a diet that differs only in the source of the protein (and thus the bioavailability of phosphorus).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* eGFR 20-45 by modified MDRD equation
* protein/creatinine ratio <5
* blood pressure <150/95
* not taking calcium binder or supplements, vitamin D, or phosphate binders
* normal serum phosphorus and calcium corrected for albumin and intact PTH <100pg/ml
* medically stable
* able to give informed consent and come for all visits

Exclusion Criteria:

* history of significant liver disease or cirrhosis
* medically unstable
* unable to tolerate diets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine if the dietary protein source affects fasting serum and urinary phosphorus excretion in patients with CKD stages 3 and 4. | 6 months after baseline

SECONDARY OUTCOMES:
To determine if the protein source affects post prandial changes in serum and urinary phosphorus in patients with CKD stages 3 and 4. | 6 months from baseline
To determine if changes in plasma FGF23 and PTH correlate with urinary phosphorus excretion in response to different protein sources in patients with CKD stages 3 and 4. | 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Moe, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Moe SM, Zidehsarai MP, Chambers MA, Jackman LA, Radcliffe JS, Trevino LL, Donahue SE, Asplin JR. Vegetarian compared with meat dietary protein source and phosphorus homeostasis in chronic kidney disease. Clin J Am Soc Nephrol. 2011 Feb;6(2):257-64. doi: 10.2215/CJN.05040610. Epub 2010 Dec 23. PMID 21183586